CLINICAL TRIAL: NCT05431634
Title: A Blinded, Randomized, Placebo-controlled, Multiple Dose Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ESK-001 Tablets Administered Over 14days to Healthy Participants
Brief Title: Multiple Dose Study to Determine Safety and Tolerability of ESK-001 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ESK-001-003
Record Dates: First submitted 2022-06-09; First posted 2022-06-24 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Safety and Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for ESK-001
  Interventions: Other: Placebo
- Experimental Drug ESK-001 (Experimental): Experimental Drug ESK-001
  Interventions: Drug: Experimental drug: ESK-001

INTERVENTIONS:
Drug: Experimental drug: ESK-001 — Multiple doses of ESK-001
  Arms: Experimental Drug ESK-001
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Multiple Dose Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ESK-001 in Healthy Participants

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

* Participant is a man or woman between the ages of 18 and 60years, inclusive, at the Screening Visit
* Participant is healthy as determined by medical history, physical examination, vital signs, and routine laboratory parameters
* Other inclusions as specified in the protocol

Exclusion Criteria:

* Participant has a prior exposure to ESK-001
* Participant has a history of hypersensitivity to any of the ingredients of ESK-001
* Other exclusions as specified in the protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 14 days
  Safety and tolerability
Incidence of Serious Adverse Events (SAEs) | Up to 14 days
  Safety and tolerability

SECONDARY OUTCOMES:
The area under plasma concentration-time curve from time zero extrapolated to last measurable concentration (AUCt) for ESK001 on Day 1 and Day 14 | Up to 14 days
  Pharmacokinetics
The area under the plasma concentration-curve over the dosing interval (AUC(0-τ)) for ESK001 on Day1 and Day 14 | Up to 14 days
  Pharmacokinetics
The observed maximum plasma concentration (Cmax) for ESK001 on Day 1 and Day 14. | Up to 14 days
  Pharmacokinetics
The time to reach the observed maximum plasma concentration (tmax) for ESK001 on Day 1 and Day 14. | Up to 14 days
  Pharmacokinetics
Apparent plasma elimination half-life (t½λz) for ESK001 on Day 1 and Day 14 | Up to 14 days
  Pharmacokinetics
Apparent clearance CL(Clearance)/F for ESK001 on Day 1 | Up to 14 days
  Pharmacokinetics
The accumulation ratio for AUC(0-τ) (RAC AUC(0-τ)) for ESK001 on Day 14 | Up to 14 days
  Pharmacokinetics
The accumulation ratio for Cmax (RAC Cmax) for ESK001 on Day 14. | Up to 14 days
  Pharmacokinetics
Cytokine induction of pSTAT expression and downstream cytokine production as a measure of tyk2 pathway inhibition by ESK001 | 14 days after first dose
  Pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bradley, Study Director — Alumis Inc
Locations (1):
- Alumis Central site, Glendale, California, United States